CLINICAL TRIAL: NCT02204709
Title: Disease Risk Reduction and n-3 Rich Rainbow Trout (Fish for Health)
Brief Title: Disease Risk Reduction and Omega-3 Rich Rainbow Trout (Fish for Health)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic & expiration of grant funds
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: GFHNRC029
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Obesity
Keywords: obese; omega-3 fatty acids; fish
MeSH Terms: conditions — Obesity | interventions — melanin-concentrating hormone gene-related peptide, tilapia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diploid Trout entrees (Experimental): Subjects will consume a 200 gram portion of 2N trout (diploid; two sets of chromosomes) twice weekly in a prepared meal.
  Interventions: Other: 2N Trout
- Triploid Trout entrees (Experimental): Subjects will consume a 200 gram portion of 3N trout (triploid; three sets of chromosomes) twice weekly in a prepared meal.
  Interventions: Other: 3N Trout
- Tilapia entrees (Experimental): Subjects will consume a 200 gram portion of tilapia twice weekly in a prepared meal.
  Interventions: Other: Tilapia

INTERVENTIONS:
Other: 2N Trout — Diploid/2N trout source
  Arms: Diploid Trout entrees
Other: 3N Trout — Triploid/3N trout source
  Arms: Triploid Trout entrees
Other: Tilapia — Tilapia/control fish source
  Arms: Tilapia entrees

SUMMARY:
The purpose of this study is to determine how eating fish raised to have different levels of omega-3 fatty acids will reduce cardiovascular risk markers in people with elevated cardiovascular risk.

DETAILED DESCRIPTION:
Consumption of fish high in long chain omega-3 fatty acids (LCn3) is associated with reduction of cardiovascular disease (CVD) risk. CVD is a major cause of death in the United States. The current obesity epidemic contributes significantly to elevated CVD risk by increasing inflammation and platelet dysfunction. Prevention of CVD is a public health goal and comprises several avenues of action, of which inclusion of LCn3-rich fish in the diet may be one of the most effective.

Obese participants will participate in a double blind, randomized, cross-over designed trial in which they will consume twice-weekly a prepared meal containing diploid (2N) farmed rainbow trout, triploid (3N) farmed rainbow trout containing higher levels of LCn3, or tilapia, a low LCn3 fish.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 30 - 39.9 kg/m2

Exclusion Criteria:

* Are allergic to fish
* Use tobacco products or nicotine in any form including snuff, pills, and patches, or e-cigarettes in the past 6 months
* Have established cardiovascular, pulmonary, and/or a metabolic disease such as diabetes
* Have uncontrolled high blood pressure
* Have alcohol, anabolic steroids, or other substance abuse issues
* Consume more than 3 alcoholic drinks/week
* Have cancer
* Are pregnant or nursing
* Take non-steroidal anti-inflammatory drugs such as aspirin, ibuprofen or Aleve, lipid modifying drugs such as statins, take medications for blood glucose such as insulin or metformin

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in platelet activation at week 6 of each treatment | Baseline, Week 6

SECONDARY OUTCOMES:
Change from baseline in plasma interleukin-6 (IL-6) at week 6 of each treatment | Baseline, Week 6
Change from baseline in plasma tumor necrosis factor alpha (TNFa) at week 6 of each treatment | Baseline, Week 6
Change from baseline in urinary prostaglandin E2 (PGE2) at week 6 of each treatment | Baseline, Week 6
Change from baseline in urinary thromboxane B2 (TxB2-M) at week 6 of each treatment | Baseline, Week 6
Change from baseline in urinary prostaglandin I2 (PGI2-M) at week 6 of each treatment | Baseline, Week 6
Change from baseline in serum thromboxane B2 (TxB2) at week 6 of each treatment | Baseline, Week 6
Change from baseline in plasma phospholipid fatty acids at week 6 of each treatment | Baseline, Week 6
Change from baseline in platelet fatty acids at week 6 of each treatment | Baseline, Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Picklo, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT02204709/ICF_000.pdf